CLINICAL TRIAL: NCT06021925
Title: Obstetrical History and Anti-HLA Antibodies Level
Acronym: OBS-HLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Etablissement Français du Sang (Nouvelle Aquitaine) (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP221333; 2021-A01199-32 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-08-25; First posted 2023-09-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Blood Donors; Anti-HLA Antibody
Keywords: Obstetrical complications; Levels of anti-HLA antibody; Chronic histiocytic intervillositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood donors tested for anti-HLA Antibody: Blood donors tested for anti-HLA Antibody between 2010 and 2020 as part of TRALI prevention program.
  Interventions: Other: Obstetrical history; Other: Anti-HLA Antibody tests

INTERVENTIONS:
Other: Obstetrical history — Selection of donors by EFS retrospectively on the basis of inclusion criteria. Information note sent by e-mail, non-opposition as well as a questionnaire to be completed online to obtain data on obstetrical history.
Other: Anti-HLA Antibody tests — Analyze responses in relation to the results of the anti-HLA Antibody tests performed at the time of donation.

SUMMARY:
Chronic histiocytic intervillositis (CHI) is associated with severe and recurrent obstetrical complications. A link between anti-HLA Antibodies (Ab) and CHI has recently been established. At the Etablissement Français du Sang (EFS), donors who have already given birth once and have high levels of anti-HLA are excluded from donating apheresis platelets and therapeutic plasma to prevent TRALI (Transfusion Related Acute Lung Injury). No studies have examined the obstetrical history of these donors. The question is: is there an association between anti-HLA levels and obstetrical complications?

DETAILED DESCRIPTION:
Chronic histiocytic intervillositis (CHI) is a rare condition with an incidence of around 5 in 10,000 pregnancies. It is defined by major infiltration of the intervillous cavity by CD68+ maternal histiocytes, associated with fibrin deposition on the villous surface.

CHI is associated with severe obstetrical complications and a very high recurrence rate, estimated at between 70% and 100%. These complications include early and late miscarriage, fetal death, severe growth retardation in surviving fetuses, and premature delivery. The survival rate reported in the literature varies between 30% and 50%.

Anti-HLA antibodies are present in 54% of pregnant women at the end of pregnancy, and their rate increases towards the end of pregnancy. The presence of HLA antibodies also increases with the number of pregnancies, and is found in up to 74% of cases after more than 2 deliveries.

The research question concerns the existence of a statistically significant association between the presence of high levels of anti-HLA antibodies and the occurrence of one or more obstetric complications.

ELIGIBILITY:
Inclusion Criteria:

* Female blood donors who have been tested for anti-HLA antibodies in the context of TRALI prevention between 2010 and 2020 at EFS Nouvelle Aquitaine [The donors meet the conditions of the Order of December 17, 2019 establishing the selection criteria for blood donors and are over 18 years old, are not protected persons and understand French well]
* Women who have already given birth at least once (non-nulliparous women)
* Women who have not expressed their opposition at the time of donation to participating in a research project and to be contacted

Exclusion Criteria:

* None [Donors meet the conditions of the Order of December 17, 2019 establishing the selection criteria for blood donors and are over 18 years old, are not protected persons and understand French well]

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Blood donors who were screened for anti-HLA Ab between 2010 and 2020 as part of TRALI prevention at the EFS Poitiers site histocompatibility laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-06-13 (Estimated); Study Completion 2024-06-13 (Estimated)

PRIMARY OUTCOMES:
To measure the association between the occurrence of obstetrical complications and the level of anti-HLA Ab measured during the screening test performed by the EFS. | 2 months
  Obstetrical complications are defined as (binomial qualitative variable) :
  * Preterm delivery < 37 WA
  * Fetal death in utero whatever the term
  * Early or late miscarriage
  * Early or late pre-eclampsia
  * Medical termination of pregnancy
  * Intrauterine growth retardation <3rd percentile

SECONDARY OUTCOMES:
Type and precocity of obstetrical complication (multinomial qualitative variable) | 2 months
  * Preterm deliveries < 37 WA and ≥ 34 WA
  * Premature deliveries < 34 WA
  * Fetal death in utero regardless of term
  * Late miscarriage < 22 WA and ≥ 14 WA
  * Early miscarriage < 14 WA
  * Late pre-eclampsia > 37 WA and ≥ 34 WA
  * Early pre-eclampsia < 34 WA
  * Medical termination of pregnancy
  * Intrauterine growth retardation <3rd percentile
Measure the association between the type and precocity of obstetrical complications according to the type of anti-HLA Ab (class I and/or class II), when these Ab are found during the screening test performed by the EFS | 2 months
  * Preterm deliveries < 37 WA and ≥ 34 WA
  * Premature deliveries < 34 WA
  * Fetal death in utero regardless of term
  * Late miscarriage < 22 WA and ≥ 14 WA
  * Early miscarriage < 14 WA
  * Late pre-eclampsia > 37 WA and ≥ 34 WA
  * Early pre-eclampsia < 34 WA
  * Medical termination of pregnancy
  * Intrauterine growth retardation <3rd percentile
Verify the absence of response bias by comparing the HLA Ab levels of responding versus non-responding donors. | 2 months
  Anti-HLA antibody rate (median)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier LAFARGE, Doctor, Principal Investigator — Etablissement Français du Sang (Nouvelle Aquitaine); Alexandra BENACHI, Professor, Study Director — APHP, Antoine Béclère Hospital, CLAMART, France
Locations (1):
- Etablissement Français du Sang Nouvelle Aquitaine, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No